CLINICAL TRIAL: NCT00913809
Title: A Two-Way Single Dose Crossover Bioequivalency of Cord's 100 mg Desipramine HCL Tablets To Merrell Dow's 100 mg Norpramin Tablets
Brief Title: To Demonstrate the Relative Bioequivalency of Cord's 100 mg Desipramine HCL Tablets To Merrell Dow's 100 mg Norpramin Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Eric Mittleberg, Ph.D, VP of Product Development, Sandoz Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 870609-D
Record Dates: First submitted 2009-06-02; First posted 2009-06-04 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2009-06

CONDITIONS: Depression
Keywords: Antidepressant
MeSH Terms: conditions — Depression | interventions — Desipramine

ARMS (2):
- 1 (Experimental): Desipramine HCL 100 mg Tablets Cord Laboratories
  Interventions: Drug: Desipramine HCL 100 mg Tablets Cord Laboratories
- 2 (Active Comparator): Norpramin 100 mg Tablets Merrell Dow Pharmaceuticals, Inc
  Interventions: Drug: Norpramin 100 mg Tablets Merrell Dow Pharmaceuticals, Inc

INTERVENTIONS:
Drug: Desipramine HCL 100 mg Tablets Cord Laboratories
  Arms: 1
Drug: Norpramin 100 mg Tablets Merrell Dow Pharmaceuticals, Inc
  Arms: 2

SUMMARY:
To demonstrate the relative bioequivalency of Cord's 100 mg Desipramine HCl tablets to Merrell Dow's 100 mg Norpramin tablets.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal finding on physical exam, medical history, or clinical laboratory results on screening.

Exclusion Criteria:

* Positive test results for HIV or hepatitis B or C.
* Treatment for drug or alcohol dependence.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 1987-12; Primary Completion 1987-12 (Actual); Study Completion 1987-12 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on AUC and Cmax | 24 days

CONTACTS AND LOCATIONS:
Overall Officials: Jules Kann, Ph.D., Principal Investigator — Biodecision Laboratories